CLINICAL TRIAL: NCT06678737
Title: CBIT+TMS R33 Phase
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: R33 phase
Record Dates: First submitted 2024-10-31; First posted 2024-11-07 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Tics; Tourette Syndrome
MeSH Terms: conditions — Tics; Tourette Syndrome

STUDY DESIGN:
Intervention Model Description: The study is a double-blinded randomized control trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Youth with chronic tics randomized to a combined treatment involving Comprehensive Behavioral Intervention for Tics (CBIT) and inhibition of the supplementary motor area (SMA) using transcranial magnetic stimulation (TMS). TMS involves theta burst stimulation (cTBS).
  Interventions: Other: CBIT +cTBS
- Control group (Sham Comparator): Youth with chronic tics randomized to CBIT and sham stimulation for TMS
  Interventions: Other: CBIT +sham cTBS

INTERVENTIONS:
Other: CBIT +cTBS — 10 daily sessions of CBIT plus cTBS, with MRI, behavioral, and clinical assessments before and after treatment and at 1-, 3-, and 6-month follow-ups.
  Arms: Experimental group
Other: CBIT +sham cTBS — 10 daily sessions of CBIT plus sham cTBS, with MRI, behavioral, and clinical assessments before and after treatment and at 1-, 3-, and 6-month follow-ups.
  Arms: Control group

SUMMARY:
Chronic tics are a disabling neuropsychiatric symptom associated with multiple child-onset mental disorders. Chronic tics affect 1-3% of youth 1 and are associated with impaired functioning, emotional and behavioral problems, physical pain, diminished quality of life, peer victimization, and a fourfold increased risk of suicide compared to the general population. Large randomized trials have demonstrated the superiority of CBIT over supportive therapy in child and adult patients. However, in these trials, only 52% of children and 38% of adults showed clinically meaningful tic improvement, meaning that 50-60% of patients do not benefit from CBIT. CBIT success relies on an ability to suppress tics that many youth lack. The central aim of CBIT is to enhance voluntary tic suppression. Better tic suppression ability drives CBIT improvement 10 and predicts lower tic burden over the course of illness. During the core CBIT procedure, competing response training, patients learn to inhibit tics by engaging in a competing motor action. However, research shows that many youth lack this fundamental tic suppression ability that CBIT aspires to enhance.

This study will examine the clinical and neural effects of a treatment combining Comprehensive Behavioral Intervention for Tics (CBIT) and transcranial magnetic stimulation (TMS) to the supplementary motor area (SMA) in young people with tic disorder.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-21 years at time of enrollment.
* Current chronic motor and/or vocal tics, defined as tics for at least 1 year without a tic-free period of more than 3 consecutive months. Tics must not be due to a medical condition or the direct physiological effects of a substance.
* At least moderate tic severity, defined as a Yale Global Tic Severity Scale total score ≥14 (≥9 for those with motor or vocal tics only).
* Full scale IQ greater than 70.
* Child, consenting parent, and adult participant required to have English fluency and literacy to ensure comprehension of study measures and instructions.
* Right-handed
* To increase external validity of findings, we will include participants taking psychotropic medications that have been stable for 6 weeks and expect to remain stable for the approximately 3-week intervention protocol (with the exception of those taking neuroleptic/antipsychotic medications). Those who previously received tic-specific therapy will be included if they meet the tic severity criterion.

Youth receiving other forms of psychotherapy will be included provided these treatments are not focused on tics. All concurrent treatments will be monitored during the study period.

Exclusion Criteria:

* Medical conditions contraindicated or associated with altered TMS risk profile, including history of intracranial pathology, epilepsy or seizure disorders, traumatic brain injury, brain tumor, stroke, implanted medical devices or metallic objects in the head, current pregnancy or girls of childbearing age not using effective contraception, or any other medical condition deemed serious or contraindicated by a study physician.
* Inability to undergo MRI (e.g., metal in body, claustrophobia, orthodontia)
* Left handedness.
* Active suicidality.
* Previous diagnosis of psychosis or cognitive disability.
* Substance abuse or dependence within the past year.
* Concurrent psychotherapy focused on tics.
* Neuroleptic/antipsychotic medications.
* Pregnant according to the medical history or a urine pregnancy test; and menstruating individuals capable of becoming pregnant and not using a highly effective form of contraception (FDA-approved hormonal contraceptive, IUD, tubal ligation)
* Taking a medication that has not reached stability criterion (same medication and dose for 6 weeks with no planned changes over the intervention period)

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2030-07-15 (Estimated); Study Completion 2030-07-15 (Estimated)

PRIMARY OUTCOMES:
Tic severity | pretreatment, 10days, 1,3,6 months
  Yale Global Tic Severity Scale, YGTSS: Gold-standard, clinician-administered tic severity scale. Includes symptom checklist of specific tic types.
Tic Suppression Task | pretreatment, 10days, 1,3,6 months
  Direct observation measure of tic suppression ability. In this paradigm, a participant is seated alone in a room in front of a computer capturing a video recording of tic occurrences for later coding by independent raters. TST will consist of two 3-min conditions: 1) free-to-tic (FT): youth is instructed to stay seated and tic freely, a measure of naturally occurring tic frequency (tics per minute); 2) suppression: youth is instructed to suppress tics. Videos will be coded to establish tic frequencies using a computerized behavioral coding program.
Tic symptoms severity | pretreatment, 10days, 1,3,6 months
  Parent/Adult Tic Questionnaire : Adult-self or parent-report measure of tic symptoms and severity
Premonitory Urge for Tics Scale | pretreatment, 10days, 1,3,6 months
  Self-report measure of intensity of urges to tic
Emotional and Behavioral functioning | pretreatment, 3,6 months
  Child/Adult Behavior Checklist: Parent- or adult-self report measuring broad emotional and behavioral functioning
Self- and parent measure of functional impairment | pretreatment, 10days, 1,3,6 months
  Patient-Reported Outcomes Measurement Information System (PROMIS-49)
Behavior Rating Inventory of Executive Function | pretreatment, 1,3,6 months
  Self- and parent-rated measure of impairment of executive function. Raw scores are converted into standardized T-scores with a mean of 50 and standard deviation of 10, higher scores reflect greater symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Conelea, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States